CLINICAL TRIAL: NCT02510391
Title: Modular Treatment for Preschool Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adam Lewin (Other)
Collaborators: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Adam Lewin, Associate Professor, University of South Florida
Organization: University of South Florida (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH-Preschool 2015
Record Dates: First submitted 2015-07-15; First posted 2015-07-29 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Anxiety
Keywords: modular; anxiety; preschool; exposure and response prevention; Cognitive behavioral therapy
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PIPA (Experimental): Modularized treatment for anxiety in children ages 3-7 years old
  Interventions: Behavioral: PIPA

INTERVENTIONS:
Behavioral: PIPA — Parent-training Intervention for Preschoolers with Anxiety (PIPA) is a behaviorally based modular treatment program for emotional and behavioral problems in young children. 12 sixty minute sessions will be delivered weekly. This intervention employs a modular format following a treatment algorithm in which therapy modules are selected by the therapist and supervisor on a session-by-session basis to address the most pressing clinical needs. Minimum session requirements for parent training/education and fear hierarchy/exposure are set to insure adequate dose of core exposure and response prevention for anxiety across cases.
  Other Names: Cognitive behavioral therapy; Exposure and response prevention; Parent training

SUMMARY:
This nonrandomized pilot study is investigating the efficacy of a modularized treatment for anxiety in children ages 3-7 years old. Eligibility is determined at a baseline assessment, followed by a second baseline assessment one month later. The treatment protocol, Parent-training Intervention for Preschoolers with Anxiety (PIPA), is flexible and allows for individualized treatments based on a treatment algorithm, ensuring that sessions address the most pressing clinical needs of each child. Treatment consists of weekly 60-minute sessions delivered over the course of 12 weeks. Symptom change is tracked weekly during brief phone assessments and a post-treatment assessment will occur following the final treatment session, approximately 12 weeks after starting treatment. Finally, all participants will complete two follow-up assessments, occurring 1-month and 6-months after the final treatment session.

DETAILED DESCRIPTION:
Early childhood mental illness is a growing public health concern, and can persist into adolescence and adulthood if left untreated. Anxiety disorders are among the most common psychiatric illnesses in preschool aged youth and place youth at significantly higher risk for anxiety, depression, substance abuse, conduct problems, and diminished academic/occupational and social/relational functioning later in life. Accordingly, there is increasing emphasis on early identification and intervention, before symptoms become entrenched to mitigate a trajectory towards longstanding impairment.

Unfortunately, empirically supported treatments for preschoolers with anxiety are limited. The few studies to date have tended to focus on relatively homogeneous samples whose symptoms resemble those in adults (e.g., worries and fears). Anxiety can present in similar ways to adult anxiety, however can also present more broadly in young children. Young children with anxiety may also present with extreme rigidity, sensory hypersensitivity, 'meltdowns'/emotional dysregulation/temper tantrums, ritualistic/routine oriented behavior, and oppositional behavior in some context. By focusing narrowly, treatments have not been adapted for the full range of anxiety presentations in early childhood.

Therefore, the proposed study evaluates a modular, parent-driven psychotherapy developed for preschool aged youth (3-7 years) with diagnostic levels of anxiety, as well as anxiety symptoms dimensionally. The treatment program, Parent-training Intervention for Preschoolers with Anxiety (PIPA), is based on empirically supported behavioral and parent-training principles as well as the investigators' recently published pilot study of preschoolers with obsessive compulsive disorder. Sixty youth will be treated during the study. PIPA focuses on exposure and response prevention therapy (E/RP) in the context of behavioral parent training, each of which have efficacy in youth with anxiety, including high functioning autism spectrum disorders (ASD). Certain parenting responses (e.g., overprotection, critical responding, accommodation of anxiety symptoms and avoidance) have been implicated in the etiology and maintenance of pediatric anxiety disorders and, in addition to E/RP, this intervention will target behavioral parent training and unhelpful parenting practices to support long-term outcomes.

In addition, this study will investigate one surrogate biomarker of anxiety in young children, fear conditioning (or more specifically, resistance to extinction). Behavioral treatment of anxiety, including the proposed PIPA intervention, relies on principles of extinction. Children and adults with anxiety disorders have been shown to have poorer fear extinction; however, there are few studies in young children examining this phenomenon. The potential to understand fear extinction in young children has implications for improving treatment efficacy and altering the negative trajectory of youth with anxiety disorders.

Eligibility will be determined at a baseline assessment. A second baseline assessment will occur one month later for those that qualify. This assessment will be used to control for symptom change due to the natural passage of time. Treatment will be delivered over 12 weeks and will include weekly 60-minute sessions. A brief phone call with an assessor each week will be used to track symptom change during treatment, and a post-treatment assessment will be conducted following the final treatment session, approximately 12 weeks later. Follow-up assessments will occur 1-month and 6-months following the final treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 7 years
* Anxiety-based concerns rated as a top problem on the Top Problems Assessment at initial assessment.

Exclusion Criteria:

* Report or evidence of severe intellectual disability or level 3 autism spectrum disorder (ASD) without accompanying intellectual/language impairment (mild ASD is not exclusionary).
* Presence of clinical features requiring a higher level of care (inpatient or partial hospital treatment).
* Unwillingness of parents to accompany their children for multiple study visits;
* Presence of a significant and/or unstable medical illness that might lead to hospitalization during the study.
* Initiation of an antidepressant within the 12 weeks preceding study enrollment, antipsychotic within 8 weeks prior to study enrollment, changes in established psychotropic medications within 8 weeks before study enrollment, or any change in alternative medications that might have behavioral effects within 6 weeks prior to study baseline assessment. Youth may remain stable on medications during the study.
* Ongoing reports of abuse/neglect or trauma reported as a primary concern.
* Extreme aggression/risk behaviors (e.g., harming animals, fire starting, violence) suggestive of conduct disorder trajectory.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-03 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety Improvement as assessed by Clinical Global Impression- Improvement (CGI-I) | Rating after the final therapy session, approximately 12 weeks after starting treatment.
  7-point clinician rating of improvement of psychopathology

SECONDARY OUTCOMES:
Key Child Problems as assessed by Top Problems Assessment (TPA) | Assess at end of treatment (approximately 12 weeks from start), 1-month following end of treatment, 6-months after completion of treatment
  obtains ratings of severity of the top three problems as identified by parent report
Child Diagnostic Presence as measured by the Schedule for Affective Disorders and Schizophrenia for School-Age Children (K-SADS) | Assess at end of treatment (approximately 12 weeks from start), 1-month following end of treatment, 6-months after completion of treatment
  Semi-structured diagnostic interview used to assess possible diagnoses via parent report
Anxiety Severity as measured by the Clinical Global Impression- Severity (CGI-S) | Assess at end of treatment (approximately 12 weeks from start), 1-month following end of treatment, 6-months after completion of treatment
  7-point clinician rating of severity of psychopathology

CONTACTS AND LOCATIONS:
Overall Officials: Adam B Lewin, Ph.D., ABPP, Principal Investigator — University of South Florida
Locations (1):
- Rothman Center for Pediatric Neuropsychiatry, St. Petersburg, Florida, United States